CLINICAL TRIAL: NCT05218239
Title: Effect of Pelvic Floor Workout on Pelvic Floor Muscle Function Recovery of Postpartum Women
Brief Title: Effect of PEFLOW on PFM Function Recovery of Postpartum Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Sun Xiuli, professor; chief physician, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH6
Record Dates: First submitted 2021-12-01; First posted 2022-02-01 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Pelvic Floor Muscle Weakness; Rehabilitation
Keywords: postpartum; global training; rehabilitation; pelvic floor muscle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine education group (Active Comparator): Routine education, including postpartum lifestyle, Kegel exercise and Knack method.
  Interventions: Behavioral: Active Comparator: Routine education group
- Global training group (Experimental): Global training was added on the basis of routine education.
  Interventions: Behavioral: Active Comparator: Routine education group; Behavioral: Experimental: Global training group

INTERVENTIONS:
Behavioral: Active Comparator: Routine education group — Behavior guidance on pelvic floor muscle function training , including Knack method education , and Kegel exercise and other pelvic floor muscle training methods were taught to postpartum women.
Behavioral: Experimental: Global training group — Global training was added on the basis of control group. The 30min-training plan is divided into 9 sections, of which, groups 1 to 8, each group takes about 3 minutes, the ninth group is cool down section, including stretching for 5 minutes and foam axis stretching for 1 minute.
  Arms: Global training group

SUMMARY:
The purpose of this study is to explore the correlation between women's pelvic floor function with their overall state of bodily functions, including body composition, physical activity levels, trunk muscle endurance, body posture, vaginal and gut microbes. The main intervention of this study is a set of global training which Includes the strength, endurance, flexibility, stability and flexibility training on the diaphragm, abdominal, lower back, as well as pelvic floor muscles, on the basis Kegel training. The primary destination of global training is to shorten the cycle of postpartum pelvic floor functional recovery, improve the effect of maternal training, and convenient in clinical promotion.

DETAILED DESCRIPTION:
Training for 2 times a week, for 12 weeks leading by a specific physiotherapist.The training intensity was evaluated by RPE self-induced fatigue scale.

ELIGIBILITY:
Inclusion Criteria:

* Newly born women within 42 days to 3 months after delivery, after the end of puerperium, initial postpartum review and pelvic floor professional outpatient screening, found that pelvic floor muscle strength decreased (Oxford Oxford muscle strength ≤ grade 3);
* Healthy before pregnancy without pregnancy complications;
* Convenient transportation, familiar with the Internet;
* Be in good condition and be able to complete the exercise program;
* Complete clinical baseline data;
* Agreed to conduct the study and signed the informed consent.

Exclusion Criteria:

* Patients with stage Ⅲ and Ⅳ pelvic organ prolapse;
* Severe urinary incontinence;
* lochia, vaginal bleeding and pregnancy;
* Serious medical diseases, such as cardiac dysfunction who wear pacemakers, neurological diseases, cognitive impairment and other pathological conditions;
* Cannot complete the intervention program;

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline pelvic floor muscle strength at 6 months or after 12 weeks training | Baseline; After 12 week training or 6th month postpartum
  The participants were instructed to contract the pelvic floor muscle correctly and allowed for one practice. Three times of maximum contraction holding for five seconds with an interval resting of five seconds were performed, and the maximum value among three was recorded as the muscle strength of maximal voluntary contraction. The result was recorded using the modified Oxford Grading scale, ranging from 0 to 5, which 0 represents no discernible pelvic floor muscle contraction and 5 represents a strong pelvic floor muscle contracion.
Change from Baseline pelvic floor electrophysiology at 6 months or after 12 weeks training | Baseline; After 12 week training or 6th month postpartum
  We use Urostym to measure pelvic floor muscle strength which can identity the strength between Type I muscle fibers and Type II muscle fibers.
Change from Baseline pelvic floor muscle strength at 1 year postpartum | Baseline; 1 year postpartum
  The participants were instructed to contract the pelvic floor muscle correctly and allowed for one practice. Three times of maximum contraction holding for five seconds with an interval resting of five seconds were performed, and the maximum value among three was recorded as the muscle strength of maximal voluntary contraction. The result was recorded using the modified Oxford Grading scale, ranging from 0 to 5, which 0 represents no discernible pelvic floor muscle contraction and 5 represents a strong pelvic floor muscle contracion.
Change from Baseline pelvic floor electrophysiology at 1 year postpartum | Baseline; 1 year postpartum
  We use Urostym to measure pelvic floor muscle strength which can identity the strength between Type I muscle fibers and Type II muscle fibers.

SECONDARY OUTCOMES:
The occurrence of SUI | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  SUI is defined by SUI symptoms or a positive result of the stress test. Before the stress test, participants are suggested to keep fully bladder. Positive result of the stress test is defined as involuntarily urinary leakage when asked to cough in the lithotomy position.
Change from Pelvic floor ultrasound indicators | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  LAM thickness, diameter of the levator hiatus and levator hiatus area
Change from Pelvic Organ Prolapse Quantitation | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  Pelvic Organ Prolapse Quantitation is measured by callipers
Change from Physical activity levels | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  We use International Physical Activity Questionnaire score to measure the overall physical activity level during postpartum period.
Change from pelvic sagittal rotation degree | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  The quantitative measurement of pelvic sagittal rotation degree on X-ray was analyzed which includes the pelvic tilt angle , the sacral slope angle, the difference of sacral slope and pelvic tilt, the ratio of the pelvic tilt angle to the sacral slope angle, the ratio of the pelvic tilt angle to the pelvic incidence angle and sacral-femoral distance.
Change from body composition | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  Body composition analysis is measured which mainly includes Body Mass Index（BMI）based on height and weight in kg/m^2.
Change from body strength | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  Hand grip strength and trunk endurance are measured to describe body strength. Hand grip strength was measured by JAMAR Plus+ grip gauge. The measurement accuracy is 0.1kg. The participants should not have visible hand defects. The grip gauge should be adjusted before measurement. When the paticipants holds the grip gauge, the second knuckle of the index finger should be at 90 degrees. At the same time, mark the best position of each hand on the grip meter. Before measurement, the participants should remove wrist jewelry to avoid injury. And the left and right hand are measured alternately for 3 times.
Change from Pelvic Floor Distress Inventory（PFDI-20）Questionnaire Score | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  The Pelvic Floor Distress Inventory Questionnaire-20 (PFDI-20) is the short-form version of the Pelvic Floor Distress Inventory (PFDI).Since it is comprised of the UDI-6, POPDI-6, and the CRADI-8, the PFDI-20 includes 20 questions.The scale scores are found individually by calculating the mean value of their corresponding questions and then multiplying by 25 to obtain a value that ranges from 0 to 100.The sum of the 3 scales are added together to get the PFDI-20 summary score, which ranges from 0 to 300.
Change from PFIQ-7 Questionnaire Score | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  The Pelvic Floor Impact Questionnaire-7 (PFIQ-7) is a shortened, less comprehensive version of the Pelvic Floor Impact Questionnaire (PFIQ).To get scale scores, the mean of each of the 3 scales is individually calculated, which ranges from 0-3, this number is then multiplied by 100 and then divided by 3.The scale scores are then added together to get the total PFIQ-7 score, which ranges from 0-300. A lower score means there is a lesser effect on quality of life.
Change from FSFI-6 Questionnaire Score | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  The 6-item Female Sexual Function Index (FSFI) is a short form of the original 19-item FSFI that measures sexual function in women.It comprises six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Desire and satisfaction items are rated on a 5-point Likert scale, ranging from 1 to 5, and the other items are rated on a 6-point Likert scale, ranging from 0 to 5. Total scores range from 2 to 30, with lower scores indicating worse sexual functioning.
Change from the Pittsburgh Sleep Quality Index (PSQI) Score | Baseline; After 12 week training or 6th month postpartum；1 year follow-up
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The 18 items consist of 7 components, and each component is scored according to the grade of 0 ~ 3. The cumulative score of each component is the total score of PSQI, and the total score range is 0~2l. The higher the score, the worse the sleep quality. It takes 5 to 10 minutes for the participants to complete the question.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Sun, PHD, Study Chair — Study Chair
Locations (1):
- The Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
(1)Date of disclosure of raw data: December 2023. Data content: original recorded data and research proposals; (2) Ways or means of sharing IPDs, contact the researchers.
Supporting Information: Study Protocol, CSR
Time Frame: 2 years
Access Criteria: contact the researchers

REFERENCES:
- [Derived] Zhu H, Zhang D, Gao L, Liu H, Di Y, Xie B, Jiao W, Sun X. Effect of Pelvic Floor Workout on Pelvic Floor Muscle Function Recovery of Postpartum Women: Protocol for a Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Sep 4;19(17):11073. doi: 10.3390/ijerph191711073. PMID 36078788